CLINICAL TRIAL: NCT02069080
Title: Imaging CXCR4 Expression in Subjects With Cancer Using 64 Cu-Plerixafor
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Lombardi Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 140050; 14-I-0050
Record Dates: First submitted 2014-02-20; First posted 2014-02-21 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07-10

CONDITIONS: Cancer
Keywords: Positron Emission Tomograhy; Metastasis
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- 1 (Experimental): All subjects are administered the study drug
  Interventions: Drug: 64-Cu-plerixafor

INTERVENTIONS:
Drug: 64-Cu-plerixafor — Five subjects with CXCR4-positive tumor sample(s) will be administered an initial intravenous (IV) infusion of 64Cu-plerixafor of up to 8+0.8 mCi (0.48+0.048 rem) not to exceed 5 g of 64Cu-plerixafor at Day 0. These subjects will undergo an initial lowdose CT scan followed by 3 consecutive torso PET scans as soon as practical after the infusion, and 2 additional PET/CT scans at 4 hours +/- 1 hour and 24 hours +/- 2 hours post-infusion. Human dosimetry will be calculated based on these results, and a maximum dose will be used, not to exceed the calculated limit of a total effective dose of 5 rem, or the radiation exposure limit for each organ.
  The remaining subjects with CXCR4-positive (n=15) and CXCR4-negative (n=5) tumor sample(s) will be administered 64Cu-plerixafor at the same or a newly calculated dose and will undergo 1 PET/CT scan between 1 and 4 hours post-infusion.

SUMMARY:
In mouse models and in patients, expression of the chemokine receptor CXCR4 on various cancers has been correlated with aggressive biological behavior, including increased rates and certain sites of metastasis, and decreased survival. Plerixafor (Mozobil ; Genzyme; Cambridge, MA) has been identified as a specific inhibitor of CXCR4, and it is currently approved by the Food and Drug Administration as a stem-cell mobilizing agent in combination with granulocyte colony-stimulating factor in the treatment of non-Hodgkin's lymphoma and multiple myeloma. Our group has recently shown that plerixafor can be labeled with the positron-emitting radionuclide copper-64((64)Cu) to form (64)Cu-plerixafor, which can be used to visualize CXCR4-positive tumor xenografts in mice using small-animal positron emission tomography (PET). Determining CXCR4 expression in tumors using (64)Cu-plerixafor and PET/computerized tomography (CT) scanning could be useful in predicting tumor behavior and responses to current and experimental therapies, including therapies targeting CXCR4, which could lead to more effective personalized cancer treatments.

This study s primary objective is to evaluate (64)Cu-plerixafor as an imaging agent for quantifying CXCR4 expression in subjects (greater than or equal to 18 years of age) with cancer; at least 1 detectable solid tumor of greater than or equal to 2 cm in diameter found outside of the lymph nodes, bone marrow, liver, gallbladder, kidney, bladder, and brain; and preexisting biopsies of the tumors obtained since the first detection of the current occurrence/recurrence of disease. The secondary objectives are to correlate (64)Cu-plerixafor standardized uptake value in the target lesion with the level of CXCR4 expression detected via immunohistochemistry and to calculate human dosimetry for (64)Cu-plerixafor.

Preexisting tumor biopsies from less than or equal to 75 subjects recruited from the National Cancer Institute and the Georgetown University Hospital will be evaluated for CXCR4 expression via immunohistochemistry. Subjects who meet the eligibility criteria will continue onto the study. Five subjects with CXCR4-positive tumor biopsies will be administered an initial intravenous infusion of (64)Cu-plerixafor (8 +/-0.8 mCi ; 0.48+/- 0.048 rem; not to exceed 5 microg of (64)Cu -plerixafor) over 2 minutes. They will then undergo an initial low-dose transmission CT scan followed by 3 consecutive torso PET scans as soon as practical after the infusion, and 2 additional PET/CT scans at 4 hours +/- 1 hour and 24 hours +/- 2 hours post-infusion. Human dosimetry will be calculated based on these results, and a maximum dose will be used, not to exceed the calculated limit of a total effective dose of 5 rem, or the radiation exposure limit for each organ. The remaining subjects with CXCR4-positive (n=15) and CXCR4-negative (n=5) tumor biopsies will be administered 64Cu-plerixafor at the same, or a newly calculated dose, and will undergo 1 PET/CT scan between 1 and 4 hours post-infusion, depending on the dosimetry results. All subjects will undergo one comprehensive final study visit between study days 19 and 23 (11-17 days after injection with (64)Cu -plerixafor). Additionally, blood will be collected 2 more times between study days 13-16 and study days 26-30 to measure blood cell counts.

...

DETAILED DESCRIPTION:
In mouse models and in patients, expression of the chemokine receptor CXCR4 on various cancers has been correlated with aggressive biological behavior, including increased rates and certain sites of metastasis, and decreased survival. Plerixafor (Mozobil ; Genzyme; Cambridge, MA) has been identified as a specific inhibitor of CXCR4, and it is currently approved by the Food and Drug Administration as a stem-cell mobilizing agent in combination with granulocyte colony-stimulating factor in the treatment of non-Hodgkin's lymphoma and multiple myeloma. Our group has recently shown that plerixafor can be labeled with the positron-emitting radionuclide copper-64(64Cu) to form 64Cu-plerixafor, which can be used to visualize CXCR4-positive tumor xenografts in mice using small-animal positron emission tomography (PET). Determining CXCR4 expression in tumors using 64Cu-plerixafor and PET/computerized tomography (CT) scanning could be useful in predicting tumor behavior and responses to current and experimental therapies, including therapies targeting CXCR4, which could lead to more effective personalized cancer treatments.

This study s primary objective is to evaluate 64Cu-plerixafor as an imaging agent for quantifying CXCR4 expression in subjects (greater than or equal to 18 years of age) with cancer; at least 1 detectable solid tumor of greater than or equal to 1.5 cm in diameter found outside of the vertebral bodies, liver, gallbladder, kidney, and bladder; and tissue sample(s) of the tumors obtained since the first detection of the current occurrence/recurrence of disease. The secondary objectives are to correlate 64Cu-plerixafor standardized uptake value in the target lesion with the level of CXCR4 expression detected via immunohistochemistry and to calculate human dosimetry for 64Cu-plerixafor.

Tumor samples from less than or equal to75 subjects recruited from the National Cancer Institute and the Georgetown University Hospital will be evaluated for CXCR4 expression via immunohistochemistry. With the exception of subjects with adrenocortical carcinoma, evaluation of tissue for expression of CXCR4 will be required before PET scanning. Subjects who meet the eligibility criteria will continue onto the study. Five subjects with adrenocortical carcinoma and/or CXCR4-positive tumor samples will be administered an initial intravenous infusion of 64Cu-plerixafor (up to 8+0.8 mCi; 0.48+0.048 rem; not to exceed 5 g 64Cu-plerixafor) at Day 0. They will then undergo an initial low-dose transmission CT scan followed by 3 consecutive torso PET scans as soon as practical after the infusion, and 2 additional PET/CT scans at 4 hours +/- 1 hour and 24 hours +/- 3 hours post-infusion. Human dosimetry will be calculated based on these results, and the dose may be adjusted, not to exceed the calculated limit of a total effective dose of 5 rem, or the radiation exposure limit for each organ. The remaining subjects will be administered 64Cu-plerixafor at the same, or a newly calculated dose, and will undergo 1 PET/CT scan between 1 and 4 hours post-infusion, depending on the dosimetry results. All subjects will undergo an assessment at the NIH or by phone on study Day 14 3. Additionally, blood will be collected 3 more times at Day 7 2, Day 14 3 and Day 21 3 to measure blood cell counts, and urine collected once more at Day 7 2.

ELIGIBILITY:
* INCLUSION CRITERIA:

Screening Phase

Subjects (greater than or equal to18 years of age) with cancer; at least 1 detectable solid tumor of greater than or equal to 1.5 cm in diameter found outside of the vertebral bodies, liver, gallbladder, kidney, and bladder; and, with the exception of adrenocortical carcinoma, preexisting tumor sample(s) of the cancer obtained since the first detection of the current occurrence/recurrence of disease are eligible to participate in the screening portion of the study.

Study Phase

Subjects of reproductive potential are eligible to enter the study if they agree to use 2 forms of contraception 3 weeks prior to the study start and 1 month after the administration of 64Cu-plerixafor, such as:

* Hormonal contraception.
* Male or female condoms with or without a spermicide.
* Diaphragm or cervical cap with a spermicide.
* Intrauterine device.

Male subjects may commence contraception beginning at the time of infusion of 64Cuplerixafor.

EXCLUSION CRITERIA:

Screening Phase

Subjects who are known to meet Study Phase exclusion criteria during the screening period may be excluded from entering the Study Phase.

Study Phase

Individuals who meet any of the following criteria are not eligible to participate in the study:

1. Karnofsky Performance Scale Index (KPSI) <70.
2. Women who are pregnant or lactating.
3. History of life-threatening cardiac arrhythmia.
4. Absolute neutrophil count <1000/microliters.
5. Platelet count <100,000/microliters.
6. Alanine transaminase, aspartate aminotransferase, alkaline phosphatase, or bilirubin levels greater than or equal to 4 times the upper limits of normal, or a calculated creatinine clearance rate of less than or equal to 50 mL/min.
7. Treatment with plerixafor or any imaging agent with a radioisotope or labeled molecule administered <10 half-lives prior to administration of 64Cu-plerixafor.
8. Research radiation exposure over the past 12 months, which if added to the radiation exposure in this study, exceeds 5 rem.
9. Allergy to plerixafor.
10. Severe claustrophobia unresponsive to anxiolytics.
11. Weight over 325 pounds.
12. History of any other illness or condition which, in the investigator s opinion, may substantially increase the risk associated with the subject s participation in the study, or may compromise the scientific objectives.

Co-Enrollment Guidelines

Co-enrollment in other trials that involve the infusion of radioactive isotopes/molecules for research purposes or plerixafor is prohibited.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-02-20; Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Uptake of 64Cu-plerixafor in the target lesion(s) of subjects expressing CXCR4 versus the uptake of 64Cu-plerixafor in the surrounding non-tumor tissues. | Two Years

SECONDARY OUTCOMES:
64Cu-plerixafor SUV in the target lesion(s) versus the level of CXCR4 expression detected via immunohistochemical staining. | Two Years
Human-absorbed doses of 64Cu-plerixafor | Six Months
The incidence and severity of adverse events (AEs) by dose group. | Two Years

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Farber, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Weiss ID, Jacobson O, Kiesewetter DO, Jacobus JP, Szajek LP, Chen X, Farber JM. Positron emission tomography imaging of tumors expressing the human chemokine receptor CXCR4 in mice with the use of 64Cu-AMD3100. Mol Imaging Biol. 2012 Feb;14(1):106-14. doi: 10.1007/s11307-010-0466-y. PMID 21347799
- [Background] Zlotnik A, Burkhardt AM, Homey B. Homeostatic chemokine receptors and organ-specific metastasis. Nat Rev Immunol. 2011 Aug 25;11(9):597-606. doi: 10.1038/nri3049. PMID 21866172
- [Background] Kang Y, Siegel PM, Shu W, Drobnjak M, Kakonen SM, Cordon-Cardo C, Guise TA, Massague J. A multigenic program mediating breast cancer metastasis to bone. Cancer Cell. 2003 Jun;3(6):537-49. doi: 10.1016/s1535-6108(03)00132-6. PMID 12842083